CLINICAL TRIAL: NCT02272153
Title: The Effects of the Combination of Egg and Whole Grains on Appetite, Blood Glucose Response and Food Intake
Brief Title: Satiety Effects of the Combination of Egg and Whole Grains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 1310M44503
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Egg refined grain (Active Comparator): Eggs with white toast
  Interventions: Other: Egg refined grain; Other: Egg Whole Grain; Other: Cereal Refined grain
- Egg whole grain (Active Comparator): Eggs with whole grain toast
  Interventions: Other: Egg refined grain; Other: Egg Whole Grain; Other: Cereal Refined grain
- Cereal Refined grain (Active Comparator): rice cereal with white toast
  Interventions: Other: Egg refined grain; Other: Egg Whole Grain; Other: Cereal Refined grain

INTERVENTIONS:
Other: Egg refined grain
Other: Egg Whole Grain
Other: Cereal Refined grain

SUMMARY:
The satiety effects of the combination of protein and fiber within egg and whole grain breakfast meals. High protein with low and high-fiber is hypothesized to be more satiating than low protein, low fiber.

DETAILED DESCRIPTION:
Subjects will consume 3 different breakfast meals. Satiety will be measured by visual analogue scales; food intake will be recorded at subsequent meal as well as 24 hour food log; blood glucose response will be assessed following test meals. Subjects will consume an ad libitum lunch meal 3.5 hours after breakfast meal and food intake will be measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy,
* non-smoking,
* BMI of 18-27,
* non-dieting,
* typically consumes breakfast/lunch

Exclusion Criteria:

* distaste for eggs,
* vegetarian,
* current smoker,
* restrained eating habits,
* recent weight change,
* history of significant disease of past medical history,
* pregnant,
* lactating irregular menstrual cycle

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Satiety | 210 minutes
  Measure satiety by visual analog scales (VAS)

SECONDARY OUTCOMES:
Food intake | 210 minutes
  ab libitum lunch provided to assess food intake variation between treatments
Blood glucose response | 180 minutes
  blood glucose response via finger stick following test meals

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Department of Food Science and Nutrition, Saint Paul, Minnesota, United States